CLINICAL TRIAL: NCT07327151
Title: Soft Rehabilitation Gloves as Assistive Technology: Enhancing Upper Limb Motor Function and Activities of Daily Living in Chronic Stroke-A Randomized Controlled Trial
Brief Title: Efficacy of Assistive Soft Gloves in Chronic Stroke Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Tugba Gokbel, Assistant Prof, MD, Kocaeli University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KAEK/16.bI.05
Record Dates: First submitted 2025-12-24; First posted 2026-01-08 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Occupational Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Soft Rehabilitation Glove (SRG) Group (Experimental): Volunteers in the research group, in addition to routine neurological rehabilitation programs, will receive rehabilitation using SRGs five days a week, totaling 15 sessions, with each session lasting 20 min.
  Interventions: Device: Sybero SRGs
- Control Group (Active Comparator): Volunteers in the control group will receive standard diagnosis/treatment protocols, including occupational therapy activities, within the same period.
  Interventions: Other: Occupational therapy

INTERVENTIONS:
Device: Sybero SRGs — Patients in this group received SRG (five days a week for a total of 15 sessions, each lasting 20 minutes) in addition to their routine neurological rehabilitation program (physiotherapy and occupational therapy). This device includes finger flexion and extension movements, grasping and releasing movements, and performing activities of daily living. Activities of daily living (such as eating, drinking, combing hair, opening jars, retrieving items from overhead shelves, carrying items, brushing teeth, and carrying bags) are determined based on the patients' functional status. The SRG is operated in passive mode, allowing finger flexion and extension movements. In mirror mode, a data glove was placed on the unaffected hand, and a SRG is placed on the affected hand. When the patient flexes their finger with the unaffected hand, signals from the data glove enables grasping of the paretic hand.
  Arms: Soft Rehabilitation Glove (SRG) Group
Other: Occupational therapy — Patients in this group received 20 min of occupational therapy (five days a week for a total of 15 sessions) in addition to their routine neurological rehabilitation program.
  Arms: Control Group

SUMMARY:
Stroke is a leading cause of disability, with hemiparesis affecting approximately 85% of survivors, particularly affecting the upper limbs, which play a critical role in the activities of daily living (ADLs). While robot-assisted rehabilitation (RAR) is gaining increasing attention owing to its capacity for intensive, repetitive, and task-specific training that promotes neuroplasticity, robot-assisted hand rehabilitation (RAHR) is not yet part of standard protocols and is understudied. This study investigated the effects of a soft rehabilitation glove (SRG) applied in addition to traditional neurorehabilitation on upper limb motor function and ADLs in individuals with chronic stroke.

DETAILED DESCRIPTION:
This study aimed to investigate the effect of SRG, used in the treatment of stroke patients, on upper limb motor functions and ADLs. Stroke, the second most common cause of death in the community after heart disease, constitutes a significant health problem leading to disability in survivors. Hemiparesis, affecting approximately 85% of post-stroke patients, specifically targets the upper limbs. This rate was observed to be 40% in patients with chronic stroke. The majority of neurological motor recovery tends to occur within the first three months and can continue for up to six months, with functional improvement being prominent in the initial six months and potentially extending for up to one year. Problems arising after stroke include muscle weakness, loss of motor control, sensory disturbances, balance impairments, contractures, and changes in muscle tone. The fundamental goal of stroke rehabilitation is to enable stroke patients to achieve the maximum possible physical, functional, and psychosocial recovery within their limitations. Due to the more complex and delicately controlled anatomical structure of the upper limbs, post-stroke prognosis significantly influences ADLs. Therefore, upper limb rehabilitation is crucial for promoting independence in ADLs and improving quality of life (QoL). The number of studies on RAR has increased rapidly over the past decade. RAR contribute to the development of neuroplasticity in the brain owing to their high intensity, repetitiveness, task specificity, interactivity, and ability to objectively evaluate patient performance. The improvements correlated with motor abilities due to this development are crucial for enhancing functional performance. According to the literature, RAHR treatments applied to stroke patients significantly contribute to the improvement of upper-limb motor functions, strength, and motor control parameters after treatment. However, RAHR therapy has not yet been included in standard diagnosis/treatment protocols for hemiplegic individuals. As it is a relatively new concept introduced in the rehabilitation environment, its use is still being explored. Current research suggests the need for further studies to determine the effects of RAHR therapy on various components of stroke rehabilitation to provide higher-quality evidence. RAR treatments have been shown to stimulate neuroplastic changes through mirror neurons and consequently facilitate widespread cortical activation, which is essential for functional recovery after a stroke. Therefore, RAHR in stroke patients can contribute to functional improvement by enabling the application of goal-oriented tasks in enriched environments and ensuring high repetitions and intensity. This study aimed to investigate the impact of SRG therapy, applied in addition to routine neurological rehabilitation programs, on the affected upper limb motor functions and ADLs in hemiplegic volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals aged 18 and above who have experienced cerebrovascular events confirmed by neuroimaging and are planned to be enrolled in a neurological rehabilitation treatment program.
2. Those whose event date was more than 3 (three) months.
3. Individuals with upper limb and hand assessment of 3 or above according to the Brunnstrom Motor Assessment Scale.
4. Those with spasticity level of 2 and below in upper limb muscle groups according the Modified Ashworth Scale.
5. Individuals scoring 24 and above on the Standardized Mini-Mental Test.

Exclusion Criteria:

1. Individuals with severe dystonia.
2. Those with severe soft tissue and/or joint contractures in the upper limbs.
3. Individuals with active reflex sympathetic dystrophy, active arthritis, fractures, circulatory disorders, or bone malignancies in the affected upper limbs.
4. Those with peripheral nerve injuries in the affected upper limb.
5. Individuals with cognitive or behavioral disorders that would hinder participation in the treatment program.
6. Those with aphasia and apraxia at a level that would hinder participation in the treatment program.
7. Individuals allergic to N Cloth and Lycra.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
Goal Assessment Scale (GAS)-Light | Post-treatment (at the end of the 3 th week)
  Functional goal attainment measurement (GAS) 5-Point Rating Scale Score Predicted Attainment (-2)Less than expected outcome (-1) Expected outcome after intervention (0)Much less than expected outcome (+1) Greater than expected outcome (+2) Much greater than expected outcome The GAS-light model is designed to assist clinicians in embedding GAS into their clinical reasoning, making GAS an integral part of the decision-making and review process, not a separate outcome measurement exercises. The fundamental differences between GAS-light and the original method are as follows: A pre-defined single scoring level, adjusted and fully documented for a zero score (i.e., a clear description of the intended level of success), all other levels are rated retrospectively. Both the individual and the treatment team are involved in both goal setting and evaluations.
Modified Frenchay Scale (MFS) | Pre-treatment and Post-treatment (at the end of 3th week)
  The MFS is a scale used to assess patients' upper limb functions and IADL (such as drawing a straight line with a ruler, opening a jar lid, fastening a clothespin, and brushing hair, etc.). This scale consists of ten activities, four unilateral and six bilateral. The MFS was used to evaluate the IADL performance of patients with stroke before and after treatment. Scoring was done for each activity as 0 (no movement), 5 (task completed), and 10 (normal movement).
Jebsen Taylor Hand Function Test | Pre-treatment and Post-treatment (at the end of 3th week)
  It is a test developed to assess the fine and gross motor functions of the hand in a standardized and objective manner. The functions of both hands were assessed using seven subtasks: writing, turning playing cards, picking up small objects, simulating eating, stacking checkers, picking up large light objects, and picking up large heavy objects. The completion time for each task was recorded separately. The tasks were performed using both hands. The test score was recorded as the time taken to complete the tasks. The seven subtasks in the test simulate activities that are commonly performed in daily life.

OTHER OUTCOMES:
Assessment of Hand and Finger Grip Strength a Hand Dynamometer | Pre-treatment and post-treatment (at the end of 3th week)
  Hand grip strength is an objective criterion for assessing the functional integrity of the upper limbs. Assessing hand grip strength provides ease and objectivity in evaluating treatment progress. The purpose of this test was to determine the maximum isometric contraction capacity of the hand and forearm muscles. A hand dynamometer was used to conduct this test. Grip strength was evaluated while the patient was sitting in a chair. The elbows should be kept close to the body and at 90-degree flexion. The wrist should be in a neutral position during this process. The individual being measured is asked to grip the dynamometer as forcefully as possible. The test results were determined by calculating the average of three measurements. Norm values for measurement: For males aged 20-69, the range is 47-40 kg, and for females, it is 30-24 kilograms.

CONTACTS AND LOCATIONS:
Locations (1):
- Kocaeli University, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Stein J. Robotics in rehabilitation: technology as destiny. Am J Phys Med Rehabil. 2012 Nov;91(11 Suppl 3):S199-203. doi: 10.1097/PHM.0b013e31826bcbbd. PMID 23080036
- [Result] Maciejasz P, Eschweiler J, Gerlach-Hahn K, Jansen-Troy A, Leonhardt S. A survey on robotic devices for upper limb rehabilitation. J Neuroeng Rehabil. 2014 Jan 9;11:3. doi: 10.1186/1743-0003-11-3. PMID 24401110
- [Result] Balasubramanian S, Klein J, Burdet E. Robot-assisted rehabilitation of hand function. Curr Opin Neurol. 2010 Dec;23(6):661-70. doi: 10.1097/WCO.0b013e32833e99a4. PMID 20852421
- [Result] Prange GB, Jannink MJ, Groothuis-Oudshoorn CG, Hermens HJ, Ijzerman MJ. Systematic review of the effect of robot-aided therapy on recovery of the hemiparetic arm after stroke. J Rehabil Res Dev. 2006 Mar-Apr;43(2):171-84. doi: 10.1682/jrrd.2005.04.0076. PMID 16847784
- [Result] Timmermans AA, Seelen HA, Willmann RD, Kingma H. Technology-assisted training of arm-hand skills in stroke: concepts on reacquisition of motor control and therapist guidelines for rehabilitation technology design. J Neuroeng Rehabil. 2009 Jan 20;6:1. doi: 10.1186/1743-0003-6-1. PMID 19154570
- [Result] Vanoglio F, Bernocchi P, Mule C, Garofali F, Mora C, Taveggia G, Scalvini S, Luisa A. Feasibility and efficacy of a robotic device for hand rehabilitation in hemiplegic stroke patients: a randomized pilot controlled study. Clin Rehabil. 2017 Mar;31(3):351-360. doi: 10.1177/0269215516642606. Epub 2016 Jul 10. PMID 27056250
- [Result] Hsieh YW, Wu CY, Liao WW, Lin KC, Wu KY, Lee CY. Effects of treatment intensity in upper limb robot-assisted therapy for chronic stroke: a pilot randomized controlled trial. Neurorehabil Neural Repair. 2011 Jul-Aug;25(6):503-11. doi: 10.1177/1545968310394871. Epub 2011 Mar 24. PMID 21436390
- [Result] Zbytniewska M, Kanzler CM, Jordan L, Salzmann C, Liepert J, Lambercy O, Gassert R. Reliable and valid robot-assisted assessments of hand proprioceptive, motor and sensorimotor impairments after stroke. J Neuroeng Rehabil. 2021 Jul 16;18(1):115. doi: 10.1186/s12984-021-00904-5. PMID 34271954
- [Result] Park S, Fraser M, Weber LM, Meeker C, Bishop L, Geller D, Stein J, Ciocarlie M. User-Driven Functional Movement Training With a Wearable Hand Robot After Stroke. IEEE Trans Neural Syst Rehabil Eng. 2020 Oct;28(10):2265-2275. doi: 10.1109/TNSRE.2020.3021691. Epub 2020 Sep 4. PMID 32886611
- [Result] Radder B, Prange-Lasonder GB, Kottink AIR, Holmberg J, Sletta K, van Dijk M, Meyer T, Melendez-Calderon A, Buurke JH, Rietman JS. Home rehabilitation supported by a wearable soft-robotic device for improving hand function in older adults: A pilot randomized controlled trial. PLoS One. 2019 Aug 6;14(8):e0220544. doi: 10.1371/journal.pone.0220544. eCollection 2019. PMID 31386685
- [Result] Liao WW, Wu CY, Hsieh YW, Lin KC, Chang WY. Effects of robot-assisted upper limb rehabilitation on daily function and real-world arm activity in patients with chronic stroke: a randomized controlled trial. Clin Rehabil. 2012 Feb;26(2):111-20. doi: 10.1177/0269215511416383. Epub 2011 Aug 12. PMID 21840917
- [Result] Villafane JH, Taveggia G, Galeri S, Bissolotti L, Mulle C, Imperio G, Valdes K, Borboni A, Negrini S. Efficacy of Short-Term Robot-Assisted Rehabilitation in Patients With Hand Paralysis After Stroke: A Randomized Clinical Trial. Hand (N Y). 2018 Jan;13(1):95-102. doi: 10.1177/1558944717692096. Epub 2017 Feb 16. PMID 28719996